CLINICAL TRIAL: NCT05287841
Title: Does the Addition of Batten Grafting Improve Nasal Outcomes in Patients Undergoing Septoplasty and Turbinate Reduction? A Pragmatic Randomized Controlled Trial
Brief Title: Does Batten Grafting Improve Nasal Outcomes in Septoplasty and Turbinate Reduction?
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 21-0204
Record Dates: First submitted 2021-05-17; First posted 2022-03-18 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Nasal Obstruction; Septal Defect; Allergic Rhinitis; Nasal Polyps; Nasal Valve Collapse
MeSH Terms: conditions — Nasal Obstruction; Heart Septal Defects; Rhinitis, Allergic; Nasal Polyps

STUDY DESIGN:
Intervention Model Description: The total number of subjects to be accrued locally is 96. We expect 96 patients to be pre-screened, enrolled (consent obtained), randomized, and complete research procedures. Each arm will have 48 patients. 48 patients in two arms for total of 96 patients.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Batten graft, plus septoplasty and inferior turbinate reduction (Experimental): In the intervention arm, a portion of the quadrangular cartilage of the nasal septum is also removed, but will be refashioned and re-implanted into the patient as an autologous batten graft. This will be performed together with standard septoplasty and turbinate reduction.
  Interventions: Procedure: Batten batten graft; Procedure: Septoplasty; Procedure: Inferior Turbinate Reduction
- Septoplasty and inferior turbinate reduction alone (Active Comparator): In the control arm, a portion of the quadrangular cartilage of the nasal septum is removed. This will be performed as a standard septoplasty and turbinate reduction.
  Interventions: Procedure: Septoplasty; Procedure: Inferior Turbinate Reduction

INTERVENTIONS:
Procedure: Batten batten graft — The batten grafts are autologous grafts from the patients' own tissue, produced from nasal septal quadrangular cartilage. This will be obtained during the septoplasty portion of the procedure. The batten graft will be used to stabilize the internal nasal valve and prevent nasal valve collapse on inspiration.
  Arms: Batten graft, plus septoplasty and inferior turbinate reduction
Procedure: Septoplasty — A portion of the quadrangular cartilage of the nasal septum is removed. This will be performed as a standard septoplasty.
Procedure: Inferior Turbinate Reduction — The bilateral inferior turbinates will be surgically ablated.

SUMMARY:
The objective of this study is to compare the effectiveness of batten grafts plus septoplasty and turbinate reduction (intervention arm) compared to septoplasty and turbinate reduction alone (control arm), both in terms of subjective and objective assessments.

DETAILED DESCRIPTION:
One of the most common reasons to pursue nasal surgery is for nasal obstruction caused by a septal deviation. Otolaryngologists frequently perform septoplasties to improve nasal obstruction due to septal deviation, leading to improved airflow and decrease office visits and medication use. Concurrently with septal deviations, the inferior turbinate tends to become hypertrophied on the contralateral side potentially causing additional nasal obstruction. While septal deviations and inferior turbinate hypertrophy are more anatomical causes of nasal obstruction, there are also other types that vary depending on nasal airflow, such as nasal valve collapse. One way to surgically correct such dynamic nasal obstruction includes alar batten grafts. These grafts are not meant to change the anatomy of the nose, but instead, function to support the weakened lateral wall. Expanding the current septoplasty procedure to include batten grafts as well as inferior turbinate reduction could possibly improve long-term outcomes, especially reducing future surgeries.

ELIGIBILITY:
Inclusion Criteria:

* Patients should satisfy all the following criteria to be considered eligible for randomization:

  1. Be age 18 or above
  2. Able to provide written informed consent
  3. Have an indication for batten graft, septoplasty and turbinate reduction according to prevailing surgical practices.

  <!-- -->

  1. Septal deviation must be present on direct or endoscopic examination
  2. Inferior turbinate hypertrophy must be present, direct examination or endoscopic examination
  3. Collapse of external nasal valve and/or lateral motion instability must be documented

  <!-- -->

  1. The ENV maye be assessed clinically by observing the alar collapse at baseline or with forced inspiration, Modified cottle may also be performed.

In all patients, endoscopic examination should document that the (a) septal deviation, (b) turbinate hypertrophy, and (c) external nasal valve collapse are the primary contributing factors of obstructed breathing.

Exclusion Criteria:

1. Septal perforation
2. History of previous functional rhinoplasty or sinus or septal surgery
3. Patients who are selected for concurrent aesthetic/cosmetic rhinoplasty
4. Untreated allergic rhinitis or allergic rhinitis unresponsive to medical management
5. Patients who have concurrent sinus surgery or polyp removal or concha bullosa resection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2021-04-30 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
Nasal Obstruction Symptom Evaluation (NOSE) score | 12 months
  1. The NOSE scale is a scoring scale from 0 to 4 (0 = no problem for quality of life, 4 = a severe problem) under 5 different parameters
  2. The sum of 5 different parameters are added up to give a range of possible sums from 0-20. This sum is then multiplied by 5 to give a final score with range 0-100.
  Ref: Stewart MG, Witsell DL, Smith TL, Weaver EM, Yueh B, Hannley MT. Development and validation of the nasal obstruction symptom evaluation (NOSE) scale. Otolaryngol Head Neck Surg 2004;130:157-163

SECONDARY OUTCOMES:
Lateral Wall Insufficiency (LWI) scores | 12 months
  Blinded, and derived by independent physician watching recorded videos 2. Grading system for lateral nasal wall collapse (0-100%). (1) Identify the junction of the upper and lower cartilages (black arrow) just above the recurvature of the lower lateral cartilage. (2) Imagine a line parallel to the nasal floor across to the septum. (3) Estimate the degree of collapse during inspiration as a percentage compared with repose.
  Ref: Tsao GJ, Fijalkowski N, Most SP. Validation of a grading system for lateral nasal wall insufficiency. Allergy Rhinol (Providence) 2013;4:e66-e68
Peak Inspiratory Flow Rate (PIFR) | 12 months
  Peak inspiratory flow rate ( PIFR ) is the maximum amount of air that can be inhaled over the time course of 1 deep breath, measured in L/min. This will be measured with a nasal spirometer.
Complications and side-effects | 12 months
  Measured using the the Common Terminology Criteria for Adverse Events (CTCAE) v5.0
  Reference https://ctep.cancer.gov/protocolDevelopment/electronic_applications/ctc.htm
Cost-effectiveness (EQ-5D-5L) | 12 month
  EQ-5D-5L is a standardized measure of health-related quality of life and validated for QALYs in rhinology research.
  Estimated total cost of each treatment arm per patient/Estimated QALY derived from EQ-5D-5L per patient = cost-per-QALY
  Reference:
  Development and preliminary testing of the new five-level version of EQ-5D (EQ-5D-5L) Herdman M, Gudex C, Lloyd A, Janssen M, Kind P, Parkin D, Bonsel G, Badia X Qual Life Res 2011 Dec;20(10):1727-1736
Reoperation incidence | 12 months
  Measured as incidence of any reoperation within study follow-up period (12 months) divided by the number of total enrollees x 100%

CONTACTS AND LOCATIONS:
Overall Officials: David Hiltzik, MD, Principal Investigator — Northwell Health
Locations (3):
- United States (3):
  - Poplar Bluff Regional Medical Center, Poplar Bluff, Missouri
  - Lenox Hill Hospital/Staten Island University Hospital, New York, New York
  - Staten Island University Hospital, Staten Island, New York